CLINICAL TRIAL: NCT00872261
Title: Adolescent Women & Microbicide Trials: Assessing the Challenges & Opportunities to Their Participation
Brief Title: Determining Characteristics and Behaviors of Adolescent Women Regarding HIV Risk and Microbicide Trial Participation
Status: Completed | Type: Observational
Sponsor: FHI 360 (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Other Study IDs: R01MH086160 (NIH); R01MH086160 (NIH); DAHBR 9A-ASPA; Tolley 1 R01 MH086160-01
Record Dates: First submitted 2009-03-30; First posted 2009-03-31 (Estimated); Last update posted 2013-05-01 (Estimated); Status verified 2013-04

CONDITIONS: HIV Infections
Keywords: Clinical Trials as Topic; Adolescent Psychology; Patient Acceptance of Health Care; HIV Risk Behaviors; Adolescents; Clinical Trial Recruitment; Microbicide Acceptability; Ethics; Mixed Methods; HIV
MeSH Terms: conditions — HIV Infections; Patient Acceptance of Health Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Proxy microbicide product: Use of vaginal lubricant as a proxy microbicide gel; use of multivitamin as proxy pre-exposure prophylaxis (PrEP) product

SUMMARY:
This study will examine characteristics and behaviors of young women in India and Tanzania to determine which challenges and opportunities exist for conducting future trials of HIV prevention treatments.

DETAILED DESCRIPTION:
HIV is an infection that damages a person's immune system and can develop into AIDS. More than 10 million women between the ages of 15 and 24 currently live with HIV or AIDS, most of them in sub-Saharan Africa and Asia. The rate of infections in women is high in part because they may not be able to use existing HIV prevention methods: remaining abstinent does not help if their partner is not also abstinent and using a male condom requires the compliance of the male. Oral and topical microbicides are products women initiate using to reduce their risk of HIV infection. Several clinical trials of these products have been conducted, but few have tested populations of young women, who may have different characteristics or behaviors from other women. This study will collect data on the characteristics and behaviors of women divided into two age groups, women age 15 to 17 and women age 18 to 21, in both Tanzania and India. This study will have four goals: (1) to determine whether and how characteristics that put women at risk for HIV differ in these age and country groups; (2) to evaluate the legal, social, cultural, and delivery factors that hinder women's participation in microbicide trials; (3) to examine the understanding and ability of women in these different groups to adhere to the requirements of clinical trial participation; and (4) to determine young women's acceptability and use of a practice gel or pill.

This study will consist of three phases. The first phase will address the first two goals by conducting repeated, in-depth interviews and discussions with a small group of sexually active adolescents in India and Tanzania, followed up by interviews with informants and relevant community members. These interviews and discussions will address differences in HIV risk characteristics between groups of women and the legal, social, cultural, and delivery factors hindering women's participation in microbicide trials. The second phase will consist of a series of workshops to define and describe a set of youth-friendly procedures for using microbicides. Community members and researchers will participate in these workshops, and some adolescents will be invited to pretest the study instruments.

The third phase will be a pilot clinical study that addresses the second two goals by asking participants to undergo evaluations over time, similar to the way they would have to in a microbicide trial. Participants will complete study visits at baseline and after 2, 4, and 6 months, during which time they will answer questions about their sexual relationships and use of risk reduction behaviors. They will also provide urine, blood, and endo-cervical swab samples for testing for pregnancy, HIV, and sexually transmitted infection. Between the 4- and 6-month visits, participants will also be asked to participate in a 2-month substudy in which they use proxy pills or gels. They will then complete interviews about their experiences using the pills or gels. Some participants who decline to participate will be invited to complete brief interviews about why they chose not to participate.

ELIGIBILITY:
Inclusion Criteria:

* Sexually active in the 3 months prior to screening
* Willing to provide biological samples and answer questions about sexual behaviors

Exclusion Criteria:

* Pregnancy
* HIV infected

Ages: 15 Years to 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Formative research will recruit adolescents and other participants from community samples in Pune, India and Dar es Salaam, Tanzania.
  Pilot clinical study will recruit adolescents from India and Tanzania through healthcare facilities, nongovernmental organizations, and other mechanisms.
Sampling Method: Non-Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2010-03; Primary Completion 2012-12 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Presence of sexually transmitted infections, such as chlamydia, gonorrhea, genital herpes, or HIV | Measured at baseline and after 4 months
Adherence to condom use | Measured over 6 months
Reasons for nonparticipation in clinical study | Measured at screening
Retention, defined as the proportion of follow-up visits during the measurement window | Measured over 6 months
Proportion of participants recruited into the microbicide substudy | Measured over 2 months

SECONDARY OUTCOMES:
Description of sexual risk patterns and psychosocial mediators of risk | Measured during formative research and during the 6-month pilot clinical study

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth E. Tolley, PhD, Principal Investigator — FHI 360; Sylvia Kaaya, PhD, Principal Investigator — Muhimbili University of Health and Allied Sciences
Locations (1):
- Muhimbili University of Health and Allied Sciences, Dar es Salaam, Tanzania

REFERENCES:
- [Derived] Tolley EE, Kaaya S, Kaale A, Minja A, Bangapi D, Kalungura H, Headley J, Baumgartner JN. Comparing patterns of sexual risk among adolescent and young women in a mixed-method study in Tanzania: implications for adolescent participation in HIV prevention trials. J Int AIDS Soc. 2014 Sep 8;17(3 Suppl 2):19149. doi: 10.7448/IAS.17.3.19149. eCollection 2014. PMID 25224611